CLINICAL TRIAL: NCT01001975
Title: Determination of Sun Protection Factors (PFA and SPF) in Sunscreen Formulas Containing Combinations of Zinc Oxide and Avobenzone
Brief Title: Determination of Sun Protection in Sunscreen Formulas (Study SR09-15)(P08236)(COMPLETED)
Acronym: PFA and SPF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18119; SR09-15; P08236 (Other: Merck)
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Results first posted 2010-12-07 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Sun Protection
Keywords: Sunscreens

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPF Testing (Experimental): Following Food and Drug Administration (FDA) guidelines for SPF testing, exposure control and product-protected site erythema responses are scored after 16 to 24 hours post-exposure to full spectrum light (Ultraviolet B radiation [UVB] and UVA).
  Interventions: Drug: Sunscreen Test Code: V53-028; Drug: Sunscreen Test Code: V53-030; Drug: Standard SPF 4 Sunscreen
- UVA Protection Testing (Experimental): Determination of Ultraviolet A Protection Factor (PFA). Following FDA guidelines, test sites exposed to UVA are scored for pigmentation responses 2 to 4 hours post-exposure.
  Interventions: Drug: Sunscreen Test Code: V53-028; Drug: Sunscreen Test Code: V53-030

INTERVENTIONS:
Drug: Sunscreen Test Code: V53-028 — Sunscreen formula containing 15% Zinc Oxide, 3% Avobenzone, and 1% Ensulizole
Drug: Sunscreen Test Code: V53-030 — Sunscreen formula containing 15% Zinc Oxide and 3% Avobenzone
Drug: Standard SPF 4 Sunscreen — 8% Homosalate Standard SPF 4 Sunscreen
  Arms: SPF Testing

SUMMARY:
Study to determine the sunscreen protection factor (SPF) and ultraviolet A protection factor (PFA) of 2 sunscreen products containing the combination of zinc oxide and avobenzone with and without ensulizole.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* Have Fitzpatrick skin types I, II, or III
* In good general health based on a medical history review
* Be free of any acute or chronic illness/disease that might interfere with or increase risk of study participation
* Be able to cooperate with the investigator and research staff
* Be willing to have the test materials applied according to the protocol
* Be capable of understanding and provide written informed consent

Exclusion Criteria:

* Subjects with a history of adverse effects upon sun exposure
* Subjects currently taking any medication that may alter the sunlight response or is a known photosensitizer
* Subjects with a history of any form of cancer, lupus, psoriasis, rosacea, porphyria cutanea tarda, connective tissue disease, diabetes or any disease that would increase the risks associated with study participation
* Subjects with an abnormal sensitivity to any sunscreen agent
* Females who indicate that they are pregnant or nursing an infant during the period of the study
* Subjects with excessive hair, blemishes, nevi, warts, moles, scars, sunburn, suntan or uneven pigmentation in the test areas
* Subjects who have been administered an investigations drug or have participated in another SPF or PFA study within 30 days prior to this study
* Subjects who are allergic to latex or latex products
* Subjects who have any conditions that would make study participation inappropriate as determined by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Sun Protection Factor (SPF) Testing: Following Food and Drug Administration (FDA) guidelines for SPF testing, exposure control and product-protected site erythema responses are scored after 16 to 24 hours post-exposure to full spectrum light (Ultraviolet Radiation A [UVA] and ultraviolet radiation B [UVB]).
Period: Overall Study
Arm/Group | Sun Protection Factor (SPF) Testing | UVA Protection Testing
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sun Protection Factor (SPF) Testing | UVA Protection Testing | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (9.8) | 38 (12.6) | 40.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Determination of Sunscreen Protection Factor (SPF)
Description: Test material (V53-028 and V53-030) and control test material (8% Homoslate SPF 4) were applied to test area. Following exposure to a series of Ultraviolet light exposures, SPF scores were recorded at 16 to 24 hours post-exposure, to determine the Minimal Erythema Dose (MED) of protected and unprotected skin. SPF was calculated as the MED of protected skin divided by the MED of unprotected skin. Expected SPF 15 is a score on a scale; range 11.34 (worst) to 19.83 (best).
Time Frame: 16 to 24 hours post-exposure
Population: Only subjects from the SPF Testing group had V53-028 and V53-030 applied for the determination of SPF
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sun Protection Factor (SPF) Testing | UVA Protection Testing
Number analyzed (Participants) | 5 | 0
Score on a scale
  V53-028 | 14.72 (2.31) |
  V53-030 | 15.00 (0.00) |

2. Primary Outcome: Determination of Ultraviolet A Protection Factor (PFA)
Description: Test materials (V53-028 and V53-030) were applied to test area. Following a series of Ultraviolet radiation A (UVA) exposures, scores were recorded at 2 and 4 hours post-exposure, to determine the Minimal Persistent Pigment-Darkening Dose (MPPD) of protected and unprotected skin. PFA was calculated as the MPPD of protected skin divided by the MPPD of unprotected skin. Expected PFA is a score on a scale; range 6.40 (worst) to 15.62 (best).
Time Frame: 2 to 4 hours post-exposure
Population: Only subjects from the UVA Protection Testing group had V53-028 and V53-030 applied for the determination of PFA
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sun Protection Factor (SPF) Testing | UVA Protection Testing
Number analyzed (Participants) | 0 | 5
Score on a scale
  V53-028 |  | 11.60 (2.01)
  V53-030 |  | 10.50 (1.12)

ADVERSE EVENTS:
Arm/Group | Sun Protection Factor (SPF) Testing | UVA Protection Testing
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that no information based on the conduct (including the protocol, the data resulting from this study or the fact that this study is being conducted) will be released without prior written consent of the sponsor, unless this requirement is superceded by the State or Federal law.